CLINICAL TRIAL: NCT07199712
Title: Ozone Therapy for the Treatment of Oral Mucositis and/or Stomatitis in Patients Undergoing Radio- and Chemotherapy in the Head and Neck District: A Prospective Clinical Trial
Brief Title: Ozone Therapy for Oral Mucositis in Patients Receiving Head and Neck Cancer Radio- and Chemotherapy
Acronym: OZOMUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-OMUC-O3
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Oral Mucositis; Oral Stomatitis; Head and Neck Cancer Squamous Cell Carcinoma; Radiotherapy Induced Mucositis; Chemotherapy Induced Mucositis
Keywords: Ozone Therapy; Oral Mucositis; Head and Neck Cancer; Chemotherapy-Induced Mucositis; Radiotherapy-Induced Mucositis; Supportive Care; Pain Management; WHO Oral Toxicity Scale; Visual Analogue Scale (VAS)
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: All enrolled patients receive the same intervention, consisting of professional in-office ozone therapy sessions combined with domiciliary use of ozonated toothpaste, mouthrinse, and gel. No control or comparator group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ozonotherapy Protocol (Professional and Home-Based) (Experimental): All participants receive professional in-office ozone therapy with the Ozono DTA device (Sweden-Martina). The first treatment is administered at baseline (T0/T1), followed by additional applications at 48 hours (T2), day 5 (T3), day 8 (T4), day 12 (T5), and day 15 (T6), if clinically indicated. In parallel, participants perform domiciliary treatment for the entire 15-day study period, consisting of daily use of an ozonated toothpaste (DentoO3, 2% ozonated sunflower oil), an ozonated mouthrinse (CollutO3, 4% ozonated sunflower oil solution), and a topical ozonated gel (Ozoral Gel, 15% ozonated sunflower oil), each applied twice daily. Clinical assessments with the WHO oral mucositis scale and the Visual Analogue Scale for pain are performed at all study visits from baseline to day 15.
  Interventions: Other: Ozone Therapy (In-Office and Home-Based Treatment)

INTERVENTIONS:
Other: Ozone Therapy (In-Office and Home-Based Treatment) — The intervention consists of professional in-office ozone therapy delivered with the Ozono DTA device (Sweden-Martina) applied to oral mucosal lesions. The first treatment is administered at baseline and additional sessions are performed at 48 hours, day 5, day 8, day 12, and day 15, if clinically required. Alongside in-office therapy, participants perform a 15-day domiciliary regimen with ozonated oral care products, including toothpaste with 2% ozonated sunflower oil, a mouthrinse with 4% ozonated sunflower oil solution, and a topical gel with 15% ozonated sunflower oil, each used twice daily. Clinical outcomes are assessed at each visit from baseline to day 15 with the WHO oral mucositis scale and the Visual Analogue Scale for pain.

SUMMARY:
Oral mucositis is a frequent and painful side effect of radio- and chemotherapy, especially in patients with head and neck cancer. It can cause severe discomfort, difficulty eating and swallowing, infections, and interruptions of cancer treatment. This study evaluates the effectiveness of ozone therapy, delivered both professionally in the dental clinic and at home with ozone-based toothpaste, mouthrinse, and gel, in reducing symptoms of oral mucositis and stomatitis.

Fifty-eight adult cancer patients with oral mucositis of at least WHO grade 1 are included. Professional ozone therapy sessions are performed in-office, combined with daily home use of ozonated products. The main goal is to determine how many days are needed for lesions to heal (WHO ≤ 1). A secondary goal is to measure pain reduction using a visual analogue scale (VAS).

This research aims to provide evidence for a supportive care protocol that may improve quality of life, reduce treatment complications, and support cancer patients during therapy.

DETAILED DESCRIPTION:
Oral mucositis and stomatitis are common toxicities in patients receiving radiotherapy, chemotherapy, or combined treatment for cancer, particularly in the head and neck region. These lesions significantly impair oral function, nutrition, and quality of life, and can lead to treatment interruptions and increased risk of infection. Current management options are limited and mainly supportive.

Ozone therapy (O₃) has demonstrated antibacterial, antifungal, antiviral, anti-inflammatory, and analgesic properties. In dentistry and oral medicine, it has been applied to promote mucosal healing, modulate inflammatory responses, and enhance local circulation. This study investigates the combined use of professional in-office ozonotherapy and domiciliary application of ozonated toothpaste, mouthrinse, and gel for the treatment of oral mucositis and/or stomatitis in cancer patients.

Fifty-eight patients are enrolled and followed over multiple time points (baseline to day 15). The primary endpoint is the time to clinical response, defined as improvement to WHO grade ≤ 1. Secondary endpoints include reduction in pain intensity assessed by the Visual Analogue Scale (VAS), as well as exploratory comparisons between patients with head and neck cancers and those with malignancies in other anatomical sites.

The trial is designed as a prospective, interventional, single-arm, open-label study. Statistical analyses will include descriptive statistics, repeated measures ANOVA or non-parametric equivalents, with significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Currently undergoing oncologic therapy (radiotherapy, chemotherapy, or combined treatment).
* Presence of oral mucositis or stomatitis of at least WHO grade 1 at baseline evaluation.

Exclusion Criteria:

* Pregnant women.
* Patients with Down syndrome.
* Patients with epilepsy.
* Patients with cardiac pacemakers.
* Patients with marked sensitivity to electrical current.
* Non-cooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Response of Oral Mucositis (WHO ≤ 1) | Baseline (initial evaluation) (T0); First treatment session (T1); 48 hours (T2; Day 5 (T3); Day 8 (T4); Day 12 (T5); Day 15 (T6).
  Clinical response is defined as the first assessment at which oral mucositis improves to WHO grade ≤ 1. Evaluations are performed at baseline (day 0) and during follow-up visits at 48 hours, day 5, day 8, day 12, and day 15. Participants who do not achieve WHO ≤ 1 by day 15 are censored at their last evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No